CLINICAL TRIAL: NCT00994695
Title: A Phase II Open and Parallel Safety, Immunogenicity and Reactogenicity Trial of Mencevax ACW135 Polysaccharide Vaccine Comparing Three Groups: 2 - 4 Year, 5 - 14 Year and 15 - 29 Year Old Ethiopians
Brief Title: Safety, Immunogenicity and Reactogenicity Trial of Mencevax ACW135 Vaccine
Acronym: ETH-TVT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Armauer Hansen Research Institute, Ethiopia (Other)
Collaborators: World Health Organization (Other); Addis Ababa University (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Dr.Ahmed Bedru Omer, One of the Principal Investigators., Armauer Hansen Research Institute
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AHRI/WHO/IVB-1
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Meningococcal Meningitis
Keywords: Trivalent meningococcal polysaccharide vaccine; Children; Safety; Immunogenicity; To assess Safety of trivalent meningococcal polysaccharide vaccine in children; To assess the immunogenicity of the trivalent polysaccharide vaccine in children
MeSH Terms: conditions — Meningitis, Meningococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: Mencevax ACW Vaccine — Mencevax ACW polysaccharide vaccine subcutaneously in the left arm at 50 μg in 0.5ml(reconstituted).
  Other Names: Mencevax ACW polysaccharide vaccine

SUMMARY:
Primary objective:

To assess the immunogenicity of the Mencevax ACW135 polysaccharide vaccine at 28 days (+6days) post vaccination in 2-4, 5-14, 15-29 year age groups and compare the immunogenicity between these age groups.

Secondary Objectives:

* To estimate the incidence of common adverse events following immunization (AEFI) of GSK Nm ACW135 polysaccharide vaccine at 1h, 1d, 2d, 3d, 7d and 28 days post-vaccination
* To assess the persistence of antibody against meningitis A, C and W135 at 11 and 23 months post vaccination in 2-4, 5-14, 15-29 year age groups

Study site:Two rural communities (Kebele) in Butajira district, Ethiopia.

Methods:

* Phase II, open and parallel safety and immunogenicity trial.
* 234 younger children (2-4 years), 145 older children (5-14 years) and 33 adults (15-29 years of age) were randomly selected from the demographic surveillance database and enrolled after screening and consenting.
* Study participant received Mencevax ACW polysaccharide vaccine 50 mg in 0.5ml subcutaneously.
* Blood samples for measuring SBA titres were collected at pre vaccination and on day 28 (+6 days) post vaccination.
* Active follow up for AEFI on post vaccination day 0, 1, 2, 3, 7, & 28.
* Primary end point was vaccine response defined as sero-conversion (in subjects initially seronegative) or a 4 fold increase (in subjects initially seropositive) in serum bactericidal antibodies (SBA) against serogroups Men A, C and W135) on post vaccination day 28. In addition seroconversion was assessed by ELISA Men A IgG on day 0 and day 28 post vaccination.
* Secondary endpoints were incidence of general and local symptoms and other adverse events following immunisation during the post vaccination period day 0 to 28 and immune persistence on post vaccination month-11 and month-23.

Results:

* No significant difference in the incidence of general or local AEFI was observed between the age groups
* The statistical analysis for the Immunogenicity data is in progress

ELIGIBILITY:
Inclusion Criteria:

1. Age between 2-29 years, both sexes, living in the selected villages of Butajira area
2. A written informed consent signed by the individual (>=18y) or caretaker/guardian (2 to 17 years of age) as 18 is the legal age of maturity in Ethiopia. Assent from children/adolescents aged 12-17 years old.
3. Free of obvious health problems ascertained by medical history and clinical examination on the day of enrolment

Exclusion Criteria:

1. Those who are unlikely to complete the follow up at 4-weeks post-vaccination.
2. Use of any investigational or non-registered drug or vaccine other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
3. Administration of blood transfusion within 2 years prior to enrolment or planned use during the study period.
4. Verbal report of previous vaccination with meningococcal serogroup A, C, Y or W135 vaccines since 1999.
5. Confirmed or suspected immunosuppressive or immunodeficient condition including HIV infection.
6. A family history of congenital or hereditary immunodeficiency.
7. History of allergic reaction to any component of the vaccine
8. Presence of any fever (defined as axillary temperature of 37.5 degree centigrade or more) and/or severe illness on the day of enrolment/ vaccination.
9. Pregnancy.
10. lactation

Ages: 2 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 412 (Actual)
Dates: Start 2005-11; Primary Completion 2006-01 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To evaluate point estimates and trends in immunogenicity after not less than 28 days (+6 days) among children 2 - 4 years as compared to children 5 - 14 years and adolescents/adults 15 - 29 years (all ages inclusive) | 28 days

SECONDARY OUTCOMES:
To assess the incidence of adverse events following vaccination at 1h, 1d, 2d, 3d, 7d and 28 days post-vaccination. | 28days
To assess the immunogenicity at 11 months and 23 months (inclusive) postvaccination. | 23 month

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Aseffa Aseffa, M.D, PhD, Principal Investigator — Senior Sientist,Deputy Director, AHRI; Ahmed Bedru Omer, M.D,Pediatrician, Principal Investigator — Clinical Trial coordinator,AHRI
Locations (1):
- Butajira Hospital, Butajīra, Southern Nationality, Ethiopia

REFERENCES:
- [Result] Aseffa A, Bedru A, Yamuah L, Arga D, Worku A, Chandramohan D, Nelson CB, Engers HD. Safety of a trivalent meningococcal ACW135 vaccine among young children in Ethiopia. Vaccine. 2007 Sep 3;25 Suppl 1:A79-82. doi: 10.1016/j.vaccine.2007.04.046. Epub 2007 May 4. PMID 17548138